CLINICAL TRIAL: NCT02957227
Title: Diagnosis of Alzheimer's Disease Using Event Related Potentials
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: VA Boston Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Katherine Turk, Neurologist, VA Boston Healthcare System
Other Study IDs: 5I01CX000736-02-COG; 5I01CX000736-02 (NIH)
Record Dates: First submitted 2016-07-29; First posted 2016-11-07 (Estimated); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Mild Cognitive Impairment
Keywords: Alzheimer's disease; Frontotemporal Dementia; Lewy Body Dementia; Diagnosis
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Frontotemporal Dementia; Lewy Body Disease; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: cohort 1: Older adults with memory impairment
  Interventions: Device: No intervention is part of this study but patients use an EEG device during observational data collection.
- 2: cohort 2: Age matched healthy controls
  Interventions: Device: No intervention is part of this study but patients use an EEG device during observational data collection.

INTERVENTIONS:
Device: No intervention is part of this study but patients use an EEG device during observational data collection.

SUMMARY:
This study evaluates the use of an EEG device using Event Related Potentials to help diagnose Alzheimer's Disease in the outpatient clinical setting.

DETAILED DESCRIPTION:
The objective of this study is to improve the accuracy of diagnosis of Alzheimer's disease in a clinic setting using an EEG device to measure event related potentials.

This study will recruit patients who are being seen with a memory complaint or the first time. It will be prospective in nature. Subjects will initially be evaluated by clinicians and then clinicians will fill out a rating questionnaire as to their level of certainty of various possible dementia diagnoses. Then, during the testing portion of the study, subjects will return to have an EEG test completed measuring event related potentials during an acoustic oddball paradigm task. The EEG will be completed by a technician who has no knowledge of the subject's clinical diagnosis. After the EEG is performed, the data will be evaluated by the study clinician in a blinded fashion. The clinician will log the EEG results as being either consistent with Alzheimer's disease or not. Finally, there will be analysis of the initial clinical rating by clinicians in comparison to a given subject's EEG results and interpretation. This will allow determination as to whether or not the clinical diagnosis was in agreement or disagreement with the EEG data and interpretation. At this time point a second clinician rating questionnaire will be completed to assess the current level of confidence and diagnostic certainty in light of the now revealed EEG data in addition to clinical data. There will also be quantitative analysis of MRI structural data regarding regional atrophy patterns as well as Amyloid PET data for some of the participants which will act as a diagnostic gold standard.

An additional aim of this study is to investigate patterns of impairment on memory testing in older adults who are malingering and reporting a memory impairment in the absence of a disorder. This aim will involve testing healthy older adults using EEG and also testing memory impaired older adults with AD and comparing the results, as well as comparing the two groups results on neuropsychologic measures of effort including the Test of Memory and Malingering (TOMM).

Impact/Significance: This proposed study could allow for increased accuracy and diagnostic certainty of the correct diagnosis among memory impaired patients and could allow for the incorporation of a new clinical technique, EEG testing among memory impaired patients.

ELIGIBILITY:
Inclusion Criteria: Cohort 1: Older adults with memory impairment: must have a physician or primary caregiver report of memory loss and must be between 50 and 100 years old.

cohort 2: Older adults who test normally on neuropsychologic testing and have no history of neurologic disorders.

Exclusion Criteria: Lack of reported memory loss by physician or primary caregiver who does not meet age limits.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a memory disorder based on caregiver or referring clinician report who are being seen in the memory disorders clinic for the first time as well as age-matched older healthy controls without a neurologic condition.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2016-07; Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Change in memory disorder diagnosis | 3 years
  The memory diagnosis will be compared between a purely clinical diagnosis and the diagnosis arrived at through use of the EEG data.

SECONDARY OUTCOMES:
EEG peak amplitude and latency | 3 years
  Will be measured in order to answer the question of whether EEG amplitude and latency are predictive of Alzheimer's disease severity, using regression analysis
Cortical, quantitative MRI volume measurements | 3 years
  MRI volumes will be assessed using quantitative MRI software to assess whether they correlate with EEG amplitude and latency data
Amyloid PET tracer uptake, Standardardized Uptake Value ratios (SUVRs) | 3 years
  Amyloid PET SUVR data will be compared to other outcome measures including EEG results and quantitative MRI as well as final clinical diagnosis.
Mini mental status exam scores | 3 years
  Quantitative results from this neuropsychological test will be used to assess level of cognitive function in subjects and will be correlated with other outcome measures.
Test of Memory and Malingering (TOMM) scores | 3 years
  TOMM scores will be compared between healthy older adults simulating a memory impairment with older adults who have AD. Also both cohorts will undergo EEG testing in order to determine if EEG along with the TOMM helps determine whether older adults are displaying true cognitive impairment, or are malingering.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Turk, MD, Principal Investigator — VA, BU
Locations (1):
- VA Boston Healthcare, Jamaica Plain, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with other investigators upon written request.